# Love Together, Parent Together (L2P2): A protocol for a feasibility study of an ultra-brief couples' relationship writing program for parents of young children

Heather Prime<sup>1\*</sup>, Amy Muise<sup>1</sup>, Veronica Benyamin<sup>1</sup>, Lehana Thabane<sup>2</sup>, Mark Wade<sup>3</sup>

<sup>1</sup>Department of Psychology, York University, 4700 Keele St, Toronto, ON M3J 1P3

<sup>2</sup>Health Research Methods, Evidence & Impact, McMaster University, 1280 Main St W,

Hamilton, ON L8S 4L8

<sup>3</sup>Applied Psychology & Human Development, University of Toronto, 252 Bloor St. West, Toronto, ON M5S1V6

\*Corresponding author: email: <a href="mailto:hprime@yorku.ca">hprime@yorku.ca</a>

Clinicaltrials.gov Registration: TBD

Other Study ID Numbers: e2021-266

Funding: Prime Family Lab at York University (generic funds)

Date (version number): November 2, 2021 (1)

#### Abstract

**Background.** The COVID-19 pandemic has introduced or amplified stress and challenge within couples' relationships. Among those who are particularly vulnerable to heightened conflict and lower relationship satisfaction during this time are interparental couples with young children, whose relationships may have already been tenuous prior to the pandemic. Stress within the interparental relationship may have ripple effects on all family subsystems and child adjustment. The Love Together Parent Together (L2P2) program is a brief, low-intensity writing intervention adapted for parents of young children that was designed to reduce conflict-related distress and prevent declines in relationship satisfaction. Based on an original writing intervention by Finkel and colleagues, L2P2 has adapted the intervention duration and study population to be appropriate to the current global context. This study examines key feasibility metrics related to this adapted program with the goal of identifying problems and informing parameters of future pilot and/or main RCTs. **Methods.** The current study is a non-randomised feasibility study, using a single-arm, pre-test/post-test design to primarily assess the feasibility of an evaluative RCT, and to secondarily assess the potential effects on outcomes to be used in a future RCT. Couples will be recruited through three community-based agencies with the goal of obtaining a sociodemographically diverse sample. The first 20 couples to enroll will be included. Baseline and post-intervention surveys will be conducted, and a writing intervention will take place (three 7minute sessions over the course of four weeks). The primary outcomes will be feasibility metrics of recruitment rates, appropriateness of eligibility criteria, sample diversity, retention, uptake, adherence, and acceptability. In addition, we will develop an objective measure of couple "weness" based on analysis of writing samples. The secondary outcomes will include couples' measures (i.e., relationship quality, perceived partner responsiveness, self-reported partner responsiveness, conflict-related distress), and additional family outcomes (i.e., parent-child relations, parental/child mental health, and parenting practices). Criteria for success are outlined and failure to meet criteria will result in adaptations to measurement schedule, intervention design, recruitment approach, and/or other elements of the program. Discussion. This feasibility study will inform several components of the procedures used for a subsequent pilot RCT, in which we will examine the feasibility of the methodology used to evaluate the program (e.g., randomization, attrition to follow up assessment/across groups, and sample size estimation, preliminary effectiveness), as well as a main RCT, which will investigate the effectiveness of the intervention on primary outcome measures and mediating pathways.

*Keywords*: Couples' relationships; Family Systems; Writing Intervention; Single-Arm Feasibility Study.

# Couples' relationships during COVID-19: Implications for young families

The COVID-19 pandemic has introduced heightened levels of stress for many couples that increase the risk of harmful dyadic processes such as decreased responsive support, hostility, and withdrawal (1). Some couples' relationships may be particularly vulnerable due to pre-pandemic stressors—namely, couples with young children. Indeed, the transition to parenthood is a challenging time, and negative changes to couples' satisfaction often persist beyond the first year postpartum (2). For instance, using a large, diverse, community sample of mothers, one study found that more than 20% of mothers reported high and worsening relationship conflict over the early childhood period (3). In the current pandemic, this developmental stage of parenthood is further threatened by distinct strains experienced by many parents. Pandemic-related stressors, including financial, family, and pandemic-specific factors have been linked to parental mental health, particularly among mothers (4), with parents reporting higher levels of depression and anxiety (5), and more frequent use of alcohol as a coping strategy compared to non-parents (6). Given the importance of individual mental health to the well-being of couples, this represents a time of acute stress to interparental relationships, which may have lasting effects.

Interparental relationships form the foundation of healthy family functioning, with strong evidence for spillover effects from the interparental relationship to other family systems (7, 8) and child adjustment (9). This may be especially true under conditions of risk (10), including stress emanating from the pandemic (11). As such, threats to the interparental relationship during this time represent a family-wide risk factor. It is therefore important to provide access to evidence-based interventions aimed to prevent the deterioration of interparental relationships during and after the pandemic, with implications for the entire family. The aim of the current study is to assess the feasibility and acceptability of an interparental intervention designed to combat declines in relationship quality amid this global crisis.

# Potential utility of a brief intervention

Prior to the pandemic, there were calls for increased translational research to inform large scale couples' interventions (12). In the current context, with widespread threat due to farreaching effects of pandemic stress, this need is even more salient. Introducing novel, brief interventions to address couples' relationships has the potential to mitigate accessibility challenges related to reach and retainment (13). One brief intervention, deemed the "Marriage Hack", targets maladaptive conflict patterns by encouraging couples to reappraise their disagreements from a neutral, third-party perspective (14). This low-resource intervention, which involves three 7-minute writing sessions (for a total of a 21-minute intervention), has been shown to buffer against normative declines in marital quality over time by reducing conflict-related distress. Such an intervention has the potential for widespread scale-up among couples at risk for relationship deterioration. In addition to its brief nature, it also has the advantage of being a fully online intervention, and will therefore reduce access barriers inherent to the pandemic and to couples with young children.

# The need for a feasibility study

The overarching goal of this research program is to evaluate the effectiveness of an adapted version of the Marriage Hack intervention with couples of young children using a randomized controlled trial (RCT), and to examine the impact of the intervention on the interparental relationship as well as other family relationships. We propose to adapt this intervention in three ways. First, the original study was conducted with a relatively low-risk sample in terms of risk for couple-related distress. The current study is considered a secondary prevention program in that we are targeting couples at risk for relationship difficulties based on developmental stage

(couples with young children) and context (a global crisis). Second, to optimize reach and retainment, we will adapt the intervention from its original 12-month course to instead run over a 6-week timeframe. The number of writing sessions will remain the same (i.e., three sessions) but will be expedited to one session every two weeks. Finally, the goal of providing this program to couples with young children is to ultimately study the cascading effects on multiple family subsystems and child adjustment. Outcomes beyond the couple relationship were not examined in the original Marriage Hack RCT.

Best practice for establishing effectiveness through an RCT requires a step-wise approach: (1) a feasibility study to address specific elements of the RCT (e.g., intervention characteristics); (2) a pilot RCT to address barriers and inform parameters of the main RCT; and (3) a main RCT to assess effectiveness (15). The current protocol describes a non-randomised, single-arm feasibility study (step 1 above), with the aim to assess feasibility, identify and rectify problems, and increase the success of a future evaluative RCT.

# **Objectives**

The primary objective of the current study is to assess the feasibility and other methodological components of the Love Together, Parent Together (L2P2) intervention to inform the parameters of a future pilot (step 2 above) and main RCT (step 3 above). L2P2 is a brief conflict reappraisal program for couples with young children designed to support whole family functioning. Primary objectives of the current feasibility study are as follows:

- (1) *Recruitment:* Establish partnership with three recruitment sources and provide examine recruitment rates to determine if additional recruitment sources are needed.
- (2) Sample: Assess whether our recruitment approach and eligibility criteria are appropriate for the intended sample (i.e., participants with mild to moderate levels of couple distress as in a secondary preventive intervention). Relatedly, we are interested in the heterogeneity of the sample obtained through this recruitment approach based on sample demographics including income/education level, racial/ethnic identification, immigration status and history, and sexual orientation/gender identity.
- (3) *Program:* Assess program retention, adherence, and uptake rates—that is, the extent to which participants complete the assessment schedule in full, engage in the three writing (intervention) sessions, and report use of conflict-reappraisal strategies in between sessions.
- (4) *Measurement:* Conduct a preliminary validation of a primary outcome measure of couple "we-ness" (16) based on a content analysis of writing samples collected during the intervention. This new measure will be used in conjunction with pre-existing self-report measures of perceived partner responsiveness and responsiveness towards one's partner for a multi-method/multi-informant assessment approach in subsequent pilot/main RCTs.
- (6) Acceptability: Examine the acceptability of the adapted intervention. We will examine whether the acceptability of the intervention varies as a function of key sociodemographic variables such as gender, race/ethnicity, and immigration status.

The secondary objective is to explore preliminary effects on couples' measures (i.e., relationship quality, perceived partner responsiveness, self-reported partner responsiveness, conflict-related distress), and other family outcomes (i.e., parent-child relations, parent/child mental health, and parenting practices) to see if the expected change is evident following participation in the intervention.

#### Methods

The current protocol is written in accordance with A guide to the reporting of protocols of pilot and feasibility trials (17), Guidelines for reporting non-randomised pilot and feasibility

studies (18) and the CONSORT extension to pilot and feasibility trials (19), with adaptations for the current non-randomised design. In addition, we have adhered to the SPIRIT guidelines for reporting protocols (completed checklist can be found in additional file 1). The current protocol was registered on clinicaltrials.gov (#XXX; Other Study ID Numbers: e2021-266), where amendments to the protocol will also be documented.

# Study design

The current study is a non-randomised feasibility study, using a single-arm, pre-test/post-test design. Couples will be recruited via three recruitment platforms via email listservs. The first 20 couples who meet eligibility criteria and consent to the research process (self-directed, online) will be included in the study. Baseline assessments will include surveys collecting information on participant sociodemographic characteristics, COVID-19 related stress, self-report measures of couples' distress, relationship quality, parenting practices, responsiveness directed towards partner, and perceived partner responsiveness, as well as the mental health of self and one target child. The intervention will take place over four weeks with three 7-minute writing intervention sessions. At the beginning of each intervention session, participants will complete a brief survey of conflict frequency, as well as use of conflict reappraisal strategies since the last session. A post-intervention survey will include all measures from baseline (except COVID-19 related stress and demographics), in addition to an acceptability survey.

# **Participants**

Eligibility criteria are as follows: (i) both participants endorse being in a relationship; (ii) partners reside in the same home; (ii) one or more children under the age of 6 living at home; (iii) both participants are over age 18 years; and (iv) both members of a couple agree to participate. Exclusion criteria included: (i) no current plans or history of separation or divorce as this is meant to be a secondary preventative intervention for couples experiencing mild-to-moderate but not severe relationship difficulties.

Recruitment sources include: (1) Moms at Work, a community, education and advocacy group supporting women in their careers; (2) Unemployed Help Centre of Windsor Inc., a nonprofit organization assisting the un/underemployed and disadvantaged person during the transition period in the reemployment process; and (3) EarlyOn Child and Family Centres, who offer free, high-quality programs for young families. These recruitment sources were selected to get a range of participants in terms of potential risk factors for relationship problems.

Listserv members from each recruitment source will receive an invitation to participate in research with a direct contact link to the L2P2 study platform via Qualtrics. Participants will go through an eligibility screen, followed by review of a letter of information and informed consent. Once participants have consented, they will be asked for their contact information and that of their partner (if they are the first member of the couple to sign up). The second member of the couple will be contacted directly by the study team via email with an invitation to enroll. Once both members of a couple have enrolled, they will be given couple and participant IDs, and a survey schedule will be set-up and executed. For a schematic diagram of the time schedule of enrolment, intervention, and assessments, see Figure 1.

#### Intervention

Given that this is a single-arm design, only an intervention group will be described. The intervention sessions will consist of two stages. First, participants will be asked to provide a "summary of a time when you and your romantic partner did not agree in the last two weeks..." focusing on "you and your partner's actions (what you said and did), not about what you were thinking or feeling." Second, participants will be asked to engage in a writing task wherein they

will be instructed to reappraise the conflict they previously reported based on the following prompts (14):

"Think about this disagreement with your partner from the perspective of a third party who wants the best for all involved. This is a person who sees things from a neutral point of view. How might this person think about the disagreement? How might this person find the good that could come from it?"

"Some people find it helpful to take this third-party perspective when they are with their romantic partner. However, almost everybody finds it hard to take this third-party perspective at all times. In your relationship with your partner, what might make it hard to take this third-party perspective, especially when you're having a disagreement with your partner?"

"Even though it is hard to take a third-party perspective, people can do it. Over the next two weeks, please try your best to take this third-party perspective when you are with your romantic partner, especially during disagreements. How might you be able to take this perspective in your interactions with your partner over the next two weeks? How might taking this perspective help you make the best of disagreements in your relationship?"

Participants will receive email reminders one week after each intervention session to prompt use of the reappraisal task. Email reminders first remind them of the prompts they wrote about during the writing session. Participants are then encouraged to use the conflict reappraisal strategy, as follows:

"As you go through your daily life, please keep in mind the benefits of adopting a third-party perspective in your romantic relationship. Sometime today (now, if the timing works), please take a few moments to think about ways you can take this point of view about conflicts in your romantic relationship."

There are no criteria for discontinuing or modifying allocated interventions. Participants will be informed that they can withdraw from participation in the study at any time and that they do not need to complete all questions in surveys or writing sessions. Participants who withdraw prematurely will be compared to completers on baseline demographic and relationship characteristics.

Several steps will be taken to improve adherence to intervention protocols. The current feasibility study will be conducted online to reduce barriers to participation. The survey and intervention sessions will be made available for mobile and/or computer users to enhance access and promote adherence. Remuneration of participants will occur as the study progresses (i.e., after each session) via email in the form of a choice of gift card. Specifically, each participant will receive \$5.00 for the baseline survey, \$10.00 for each of the three intervention sessions, and \$5.00 for the post-intervention survey (\$40.00 per participant for full participation). Reminders of study timelines and survey/intervention session expiry dates will be provided by email.

## **Outcomes and Analysis**

Table 1 presents all study objectives with associated outcomes, and criteria for success of feasibility, hypothesis for secondary outcomes, and methods of analyses, when applicable. Feasibility outcomes will be reported descriptively using descriptive statistics, means (standard deviations) and frequencies/percentages. Analyses for pre-post change and validation of an objective primary outcome measure are described in Table 1. If success indicators are not met, we will make changes to study design accordingly (e.g., expand recruitment sources, adjust eligibility criteria, adapt intervention schedule and/or compensation). Analyses will include all

participants who complete baseline assessments, using Bayes estimation, which is more robust with small sample sizes.

# Sample size:

We chose the sample size of 20 couples (with expected attrition), with the goal of having data for 15 couples (N = 30). This will allow us to examine rates of recruitment over several weeks, appropriateness of eligibility criteria and reasons for exclusion, diversity of sample, retention, adherence, and uptake, as well as preliminary analyses examining pre-post change and the validity of a new primary outcome measure.

The current protocol does not include stopping or discontinuing guidelines.

# Data Management

No data entry is required as participants provide responses directly into Qualtrics. Study protocols have been developed by the Principal Investigator (PI: first author) which outline clear steps for enrolling study participants and scheduling surveys and compensation schedules. Data quality checks will be conducted at regular check points throughout data collection by the PI. Steps will be taken to ensure linking of participants within couples and over time and independent completion of surveys. Embedded data will be used across surveys to ensure consistency in reporting on specific children. Range checks will be conducted on all data to ensure valid values.

#### Ethics and dissemination

Ethics approval has been granted by York University (Certificate #: e2021-266). Changes to the protocol will be reported in the publication of study findings. Informed consent will be completed online (see additional file 2).

All information provided by participants will be kept private and confidential. An electronic file linking participant contact information with their couple identification numbers will be only accessible by the PI (first author) and research coordinator. Qualtrics servers will contain email addresses linked to each participant's data to allow for communication with participants (i.e., sending out reminders and surveys). Any data shared with the research team will contain only the participant codes, and will be securely transferred using an encrypted email or secure server.

All study data will be temporarily stored on Qualtrics before anonymized records are sent to York University secure servers (OneDrive). Qualtrics is protected by high-end firewall systems. Qualtrics uses Transport Layer Security (TLS) encryption (also known as HTTPS) for all transmitted data. Anonymized data will be made available to the senior investigators (first, second, and senior authors), and their research assistants and students (current and future) under the direct supervision of the research team.

We will destroy any personally-identifiable data at the end of the study. We will keep non-identifiable data to comply with open science and data sharing practices, as well as to allow for future analysis of data.

Dissemination plans include traditional outlets (e.g., peer-review journals and conferences), and sharing with the general public through social media and community talks (in conjunction with recruitment partners). American Psychological Association 'Publication Practices and Responsible Authorship' guidelines will be used to determine authorship.

#### Discussion

The main objectives of the current feasibility study are to examine the feasibility, acceptability, and practicality of an adapted intervention designed for couples with young children. Considerations relate to processes, resources, and scientific factors such as recruitment rates, appropriateness of eligibility criteria and sample diversity, retention, adherence, and

uptake, primary outcome measure development, and preliminary examination of change in outcome measures. We will also conduct a participant survey to assess acceptability of the intervention program, stratified by subgroups.

Findings will inform the parameters and research protocol of a future pilot RCT, the aim of which will be to assess the feasibility of examining the effectiveness of the intervention program in a subsequent main RCT. Specifically, we expect the results of this feasibility study to inform whether a future pilot RCT will be planned and what changes may need to occur, if any, prior to executing the pilot RCT.

With appropriate adaptations, the "wise intervention" presented by Finkel and colleagues (2013) has the potential to meet a pressing need for a widescale program to prevent the sequelae of the COVID-19 pandemic on interparental relationships, family functioning, and child adjustment. The current feasibility study is a critical first step to ensuring successful implementation of future pilot and main RCTs that will investigate the effectiveness of using this intervention with a new population (couples with young children) and in the context of an ongoing pandemic, and its aftermath.

#### **Declarations**

# Ethics approval and consent to participate

Ethics approval has been granted by the Office of Research Ethics at York University (Certificate #: e2021-266).

# **Consent for publication**

Not Applicable

# Availability of data and materials

Not Applicable

# **Competing interests**

The authors declare that they have no competing interests.

#### **Funding**

The current feasibility study is funded by York University, Faculty of Health, with generic funds provided to the Principal Investigator (H. Prime). Funders have no role in the project, including in study design, collection, management, analysis, and interpretation of data, writing of the report, and/or decision to submit the report for publication.

#### **Authors' contributions**

HP: Study conceptualization and design, oversight of the development of the study protocol, survey development, recruitment, and data collection, initial draft of the manuscript.

AM: Study conceptualization and design, substantive revision of the manuscript.

VB: Development of the study protocol, survey development, and substantive contributions to the drafting of the manuscript.

LT: Study conceptualization and design, substantive revision of the manuscript.

MW: Study conceptualization and design, substantive revision of the manuscript.

All authors have approved the submitted version of the manuscript and have agreed to be personally accountable for their contributions.

#### Acknowledgements

Thank you to Drs. Dillon Browne, Karen Fergus, and Eli Finkel, for their consultation on study design. In addition, thank you to Gillian Shoychet for critically reviewing the study protocol and survey development, and to Alexandra Markwell for her coordination of the project.

## **Authors' information (optional)**

Not applicable.

# **Tables**

# Table 1

| Table 1 | | | |
|---|---|---|---|
| Primary Objectives To Determine: | Outcome | Criteria for 'success' of feasibility/hypothesis | Method of analysis |
| Recruitment | Number of participants Accessed (I.e., initiate registration) per week, stratified by recruitment source | 10 couples per week over<br>the course of 4 weeks who<br>access our registration site | Descriptive statistics |
| | Number of participants Enrolled per week, stratified by recruitment source | 5 couples per week over the course of 4 weeks who enroll in the study | |
| Eligibility<br>criteria | % interested participants that<br>meet <i>Inclusion Criteria</i> (with<br>reasons for exclusion) | < 50% of participants are excluded for any one criterion. | |
| Sample diversity | % participants income <= regional median, <= high school degree | > 30% of our sample has 1+ indicator. | |
| Sample diversity (race/ethnicity/immigration) | % participants racialized, immigrant | > 30% of our sample has 1+ indicator. | |
| Sample<br>diversity<br>(sexual<br>orientation/<br>gender) | % participants non-<br>heterosexual, gender non-<br>conforming | > 30% of our sample has 1+ indicator. | |
| Mild-moderate<br>risk for<br>relationship<br>distress | % participants scoring 'clinical' (>13) on the <i>Dyadic Adjustment Scale</i> (20) % participants scoring 'high' (>29) on the <i>COVID-19 Family Stressor Scale (21)</i> | < 50% of eligible participants. | |
| Participant retention | % participants who remain in<br>study until end of post-<br>intervention assessment | > 90% of participants | |
| Participant adherence | % participants who complete 2/3 intervention sessions | > 90% of participants | |
| Participant uptake | % participants reporting some use of conflict reappraisal outside of sessions | > 80% of participants | |
| Acceptability | % of participants reporting at least 'good' on 80 % or more indicators on an <i>Implementation Acceptability Scale</i> assessing attitude, burden, perceived effectiveness, and ethicality (22). | > 80% of participants,<br>(stratified by gender,<br>immigrant status, and<br>racialized groups) | |

| Primary | Objective assessment of we- | Inter-rater reliability | |
|---|---|---|---|
| outcome | ness (16) based on content | (Cronbach's alpha > .80) | |
| measure | analysis of writing samples. | Internal consistency | |
| development | Will include an analysis of first- | (Cronbach's alpha > .70) | |
| | person plural pronouns (we, us, | Significant group | |
| | our, ours), reference to partners' | differences between male | |
| | internal states (beliefs, desires, | and female participants | |
| | intentions), and positive | based on t-tests ( $p < .05$ ) | |
| | affective language (23) | Significant correlations ( $p <$ | |
| | | .05) with indices of | |
| | | convergent validity (i.e., | |
| | | self-reported responsiveness, | |
| | | partner reported perceived | |
| | | partner responsiveness). | |
| Secondary | Couples' Relationship Quality: | Intervention will improve | 3-level multilevel models, |
| objective | Perceived Relationship Quality | outcomes from baseline to | similar to regression analysis |
| To Explore: | Scale (24) | post-intervention surveys | but accounting for clustering |
| | Conflict-Related Negativity: | post intervention surveys | within data structure |
| Pre-Post | two items following fact-based | | Within data structure |
| Change in | summary: "I was angry at my | | |
| Outcome | partner for his/her behavior | | |
| Measures | during this conflict," "My | | |
| | partner's behavior during this | | |
| | conflict was highly upsetting to | | |
| | me" (14). | | |
| | Perceived Partner | | |
| | Responsiveness/Responsiveness Directed Towards Partner: | | |
| | Two eight-item scales will | | |
| | assess participants' perceptions | | |
| | of their partners | | |
| | responsiveness/insensitivity and | | |
| | their own | | |
| | responsiveness/insensitivity | | |
| | towards their partner, | | |
| | respectively (25) | | |
| | Parent-Child Relations, | | |
| | Parenting Practices Scale from | | |
| | the Ontario Child Health Study | | |
| | Parant Mantal Health V10 | | |
| | Parent Mental Health, K10<br>Psychological Distress Scale | | |
| | (27) | | |
| | Child Emotional and | | |
| | Behavioural Problems, | | |
| | Pediatric Symptom Checklist | | |
| | (Baby, Preschool, and Standard | | |
| | versions) (28) | | |

# **Figures**

Figure 1
Schedule of enrolment, intervention, and assessments.

| Schedule of emolinem, | sintervention, and assessments. Study Period | | | | | |
|---|---|---|---|---|---|---|
| | Enrolment | <u> </u> | | | | |
| TIMEPOINT | -t <sub>1</sub> | t₁<br>Week 0 | t <sub>2</sub> Week 1 | t <sub>3</sub><br>Week 3 | nt<br>t₄<br>Week 5 | t₅<br>Week 6 |
| ENROLMENT: | | | | | | |
| Eligibility screen | Х | | | | | |
| Informed consent | Х | | | | | |
| Contact Information | X | | | | | |
| Allocation | | | | | | |
| INTERVENTIONS: | | | | | | |
| [Intervention A] | | | Х | Х | Х | |
| ASSESSMENTS: | | | | | | |
| Demographics,<br>COVID-19 Stress,<br>Relationship Distress | | Х | | | | |
| Couples' relationship quality, perceived partner responsiveness, responsiveness to partner, parent mental health, child mental health, parent-child relations | | Х | | | | X |
| Conflict-Related<br>Negativity | | | Х | Х | Х | |
| Use of Conflict<br>Reappraisal Strategy | | | | X | Х | |
| Acceptability | | | | | | Χ |

#### References

- 1. Pietromonaco PR, Overall NC. Applying relationship science to evaluate how the COVID-19 pandemic may impact couples' relationships. American Psychologist. 2020;76(3):438-450.
- 2. Kluwer ES. From partnership to parenthood: A review of marital change across the transition to parenthood. Journal of Family Theory & Review. 2010;2(2):105-25.
- 3. Madigan S, Plamondon A, Jenkins JM. Marital conflict trajectories and associations with children's disruptive behavior. Journal of Marriage and Family. 2017;79(2):437-50.
- 4. Wade M, Prime H, Johnson D, May SS, Jenkins JM, Browne DT. The disparate impact of COVID-19 on the mental health of female and male caregivers. Social Science & Medicine. 2021;275:113801.
- 5. COVID-19 national survey dashboard https://www.camh.ca/en/health-info/mental-health-and-covid-19/covid-19-national-survey2020
- 6. Wardell JD, Kempe T, Rapinda KK, Single A, Bilevicius E, Frohlich JR, et al. Drinking to Cope During COVID-19 Pandemic: The Role of External and Internal Factors in Coping Motive Pathways to Alcohol Use, Solitary Drinking, and Alcohol Problems. Alcoholism: Clinical and Experimental Research. 2020;44(10):2073-83.
- 7. Krishnakumar A, Buehler C. Interparental conflict and parenting behaviors: A meta-analytic review. Family relations. 2000;49(1):25-44.
- 8. Kitzmann KM. Effects of marital conflict on subsequent triadic family interactions and parenting. Developmental psychology. 2000;36(1):3-13.
- 9. Buehler C, Anthony C, Krishnakumar A, Stone G, Gerard J, Pemberton S. Interparental conflict and youth problem behaviors: A meta-analysis. Journal of Child and family studies. 1997;6(2):233-47.
- 10. Masarik AS, Conger RD. Stress and child development: A review of the Family Stress Model. Current Opinion in Psychology. 2017;13:85-90.
- 11. Prime H, Wade M, Browne DT. Risk and resilience in family well-being during the COVID-19 pandemic. American Psychologist. 2020;75(5):631-43.
- 12. Pietromonaco PR, Collins NL. Interpersonal mechanisms linking close relationships to health. American Psychologist. 2017;72(6):531-42.
- 13. Kanter JB, Schramm DG. Brief interventions for couples: an integrative review. Family Relations. 2018;67(2):211-26.
- 14. Finkel EJ, Slotter EB, Luchies LB, Walton GM, Gross JJ. A brief intervention to promote conflict reappraisal preserves marital quality over time. Psychological Science. 2013;24(8):1595-601.
- 15. Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Bmj. 2008;337:a1655.
- 16. Fergus K. Theoretical and methodological underpinnings of resilience in couples: Locating the 'We'. Couple Resilience: Springer; 2015. p. 23-42.
- 17. Thabane L, Lancaster G. A guide to the reporting of protocols of pilot and feasibility trials. Springer; 2019;5(1).
- 18. Lancaster G, Thabane L. Guidelines for reporting non-randomised pilot and feasibility studies. Pilot and Feasibility Studies. 2019;5(1).
- 19. Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, et al. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016;:i5239.

- 20. Sabourin S, Valois P, Lussier Y. Development and validation of a brief version of the dyadic adjustment scale with a nonparametric item analysis model. Psychological assessment. 2005;17(1):15-27
- 21. Prime H, Wade M, May SS, Jenkins JM, Browne DT. The COVID-19 Family Stressor Scale: validation and measurement invariance in female and male caregivers. Frontiers in Psychiatry. 2021;12.
- 22. Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC health services research. 2017;17(1).
- 23. Allgood SM, Seedall RB, Williams RB. Expressive writing and marital satisfaction: a writing sample analysis. Family Relations. 2020;69(2):380-91.
- 24. Fletcher GJ, Simpson JA, Thomas G. The measurement of perceived relationship quality components: A confirmatory factor analytic approach. Personality and Social Psychology Bulletin. 2000;26(3):340-54.
- 25. Crasta D, Rogge RD, Maniaci MR, Reis HT. Toward an optimized measure of perceived partner responsiveness: Development and validation of the perceived responsiveness and insensitivity scale. Psychological Assessment. 2021;33(4):338-55.
- 26. Boyle MH, Georgiades K, Duncan L, Comeau J, Wang L, Team OCHS. The 2014 Ontario child health study—methodology. The Canadian Journal of Psychiatry. 2019;64(4):237-45.
- 27. Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek D, Normand S et al. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychological medicine. 2002;32(6):959-76.
- 28. Murphy JM, Bergmann P, Chiang C, Sturner R, Howard B, Abel MR, et al. The PSC-17: subscale scores, reliability, and factor structure in a new national sample. Pediatrics. 2016;138(3).